CLINICAL TRIAL: NCT06917508
Title: A Non-Randomized, Multiple-Dose, Open-Label, Single Sequence Study to Evaluate the Effect of Concomitant Administration of EDP-323 on the Pharmacokinetics and Safety of Midazolam, Caffeine, and Rosuvastatin in Healthy Participants
Brief Title: A Study to Evaluate the Drug-Drug Interaction of EDP-323 With Midazolam, Caffeine, and Rosuvastatin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EDP 323-006
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: RSV Infection; Drug Drug Interaction
Keywords: Drug Drug Interaction
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Midazolam; Caffeine; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- EDP-323, midazolam, caffeine and rosuvastatin (Experimental): Subjects will receive EDP-323, midazolam, caffeine and rosuvastatin throughout the treatment period on respective dosing days
  Interventions: Drug: EDP-323; Drug: Midazolam; Drug: Caffeine; Drug: Rosuvastatin

INTERVENTIONS:
Drug: EDP-323 — Subjects will receive EDP-323 once daily on Days 5-15
Drug: Midazolam — Subjects will receive midazolam once daily on Days 1 and 12
Drug: Caffeine — Subjects will receive caffeine once daily on Days 1 and 12
Drug: Rosuvastatin — Subjects will receive rosuvastatin once daily on Days 2 and 13

SUMMARY:
The primary aim of this study is to assess the effect of EDP-323 on the pharmacokinetics and safety of midazolam, caffeine, and rosuvastatin in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 65 years, inclusive
* Screening body weight >50 kg and body mass index (BMI) of 18 to 32 kg/m2
* Female subjects of childbearing potential must agree to use two effective methods of contraception from the date of Screening until 30 days after the last dose of EDP-323. A male participant who has not had a vasectomy and is sexually active with a woman of childbearing potential must agree to use effective contraception from the date of Screening to 90 days after his last dose of study drug.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease
* Pregnant or nursing females
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy)
* Positive for HIV or hepatitis
* Positive urine drug screen
* Current tobacco smokers or use of tobacco within 3 months prior to Screening.
* Received any vaccine, an investigational agent, or biological product within 28 days or 5 times the t½ of receipt of study drug, whichever is longer.
* Drug sensitivity to midazolam, caffeine, rosuvastatin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Cmax of midazolam, caffeine, and rosuvastatin with and without the coadministration of EDP-323 | Up to 17 Days
AUC of midazolam, caffeine, and rosuvastatin with and without the coadministration of EDP-323 | Up to 17 Days

SECONDARY OUTCOMES:
Safety measured by adverse events | Up to 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- ICON, plc, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No